CLINICAL TRIAL: NCT01248650
Title: A Clinical Study to Investigate Pharmacokinetics and Safety of Single-Dose TRK-820 Soft Capsule in Patient With Hemodialysis
Brief Title: Safety Study of TRK-820 for Patient With Hemodialysis
Acronym: TRK-820
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Collaborators: Toray Industries, Inc (Industry)
Responsible Party: Hogan Park, SK Chemicals Co.,Ltd.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRK-820_HD_I_2008
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Chronic Renal Failure
Keywords: Safety evaluation; Pharmacokinetic analysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — TRK 820

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRK-820 5 μg (Active Comparator): Taking TRK-820 5μg(two 2.5μg soft capsules) once on the first day of hospitalization by oral route
  Interventions: Drug: nalfurafine hydrochloride
- TRK-820 2.5μg (Active Comparator): Taking TRK-820 2.5μg(one 2.5μg soft capsule) once on the first day of hospitalization by oral route
  Interventions: Drug: nalfurafine hydrochloride

INTERVENTIONS:
Drug: nalfurafine hydrochloride

SUMMARY:
The purpose of this study is to observe pharmacokinetics and safety of nalfurafine hydrochloride in patients receiving hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic renal failure who receive dialysis three times a week on a regular basis and do not expect an important change in treatment nor a rapid change in conditions
* Patients aged 20 years or older
* Patients whose post-dialysis BMI measured at the nearest time before the singing day is in the range of 70 ~ 130 %
* Patients who can understand and follow instructions and participate in the study during the entire study period
* Patients who signed the informed consent form before participating in the study

Exclusion Criteria:

* Patients who have confirmed malignant tumor
* Patients with cognitive impairment including depression, schizophrenia and dementia
* Patients with hepatic cirrhosis as a complication
* Patients with drug allergy to opioids
* Patients with drug dependency or allergic disease (including skin response to UV radiation)
* Patients who participated in other study and received the investigational drug within 1 month before the signing day
* Patients who participated in other TRK-820 study within 4 weeks before the signing day
* Pregnant or lactating women or premenopausal women of childbearing potential who do not conduct contraception
* Patients who received any of the following drugs within 2 weeks before Day 1

  1. Azole antifungal agents

     1. Ketoconazole
     2. Fluconazole
     3. Itraconazole
     4. Clotrimazole
  2. Macrolide antibiotics

     1. Erythromycin
     2. Midecamycin
     3. Josamycin
     4. Roxithromycin
     5. Clarithromycin
     6. Triacetyloleandomycin
  3. Ritonavir
  4. Cyclosporine
  5. Nifedipine
  6. Cimetidine
  7. Amiodarone
* Patients who had the following drinks and foods within 2 weeks before Day 1

  1. Foods and drinks containing grape fruit juice
  2. Food and drinks containing St. John's wort
* Patients who participated in other clinical study during the period between the singing day and hospitalization (Day 1)
* Patients who smoked and drank from three months before the signing day
* Patients who are ineligible for the clinical study for other reasons at the investigator's discretion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wooseong Huh, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea